CLINICAL TRIAL: NCT03579849
Title: Pulmonary Perfusion by Iodine Subtraction Mapping CT Angiography in Acute Pulmonary Embolism: a Diagnostic Accuracy Study Versus Pulmonary Perfusion SPECT.
Brief Title: Pulmonary Perfusion by Iodine Subtraction Mapping CT Angiography in Acute Pulmonary Embolism
Acronym: PASEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC18.0083 (PASEP)
Record Dates: First submitted 2018-06-11; First posted 2018-07-09 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perfusion SPECT (Experimental): Included patients with a diagnosis of acute PE on CTPA and who had a subtraction iodine mapping CT will undergo a SPECT/CT within 24 hours.
  Each lung subtraction iodine mapping CT will be interpreted blindly by 3 radiologists. Each of the 20 lung segments will be interpreted as normoperfused or hypoperfused.
  Each perfusion SPECT will be interpreted blindly by 3 nuclear medicine physicians. Each of the 20 lung segments will be interpreted as normoperfused or hypoperfused.
  Interventions: Diagnostic Test: Pulmonary tomoscintigraphy

INTERVENTIONS:
Diagnostic Test: Pulmonary tomoscintigraphy — The included patients will benefit from pulmonary tomoscintigraphy within 24 hours after the diagnosis of pulmonary embolism. Each tomoscintigraphy will be interpreted blindly by 3 nuclear physicians. Each of the 20 lung segments will be interpreted as normoperfused or hypoperfused.

SUMMARY:
* Pulmonary embolism (PE) is a diagnostic and therapeutic challenge. The risk of death of untreated PE is approximately 25%. On the other hand, anticoagulant treatment is associated with a haemorrhagic risk (2% of major haemorrhagic accidents per year, of which 10% are fatal). A diagnostic accuracy is therefore necessary.
* Two approaches are available to diagnose PE:

  1. A functional approach, represented by pulmonary ventilation / perfusion scintigraphy (V / P), which looks for the functional consequences of PE. The main disadvantage of this approach is that there is a high rate of non-diagnostic examinations. On the other hand, it allows a mapping of pulmonary perfusion at the microcapillary scale, and thus allows the quantification of the vascular obstruction index, which would be an independent risk factor of PE recurrence.
  2. A morphological approach, represented by CT pulmonary angiography (CTPA), which allows the visualisation of the clot itself. This approach is currently the most used but has some limitations, including a risk of over-diagnosis of pulmonary embolism and the inability to reliably quantify the index of vascular obstruction.

Lung subtraction iodine mapping CT is a new technique allowing, during the realization of a CTPA, without additional irradiation, to provide a mapping of the iodine. This mapping of iodine could potentially be used to evaluate pulmonary perfusion.

It would then be possible to obtain, during a single examination, in addition to the anatomical information of the thoracic angioscan, information on the pulmonary perfusion and thus to assess the functional consequences of PE.

No study to date has evaluated the performance of the pulmonary subtraction CT for the evaluation of pulmonary perfusion in the context of acute pulmonary embolism suspicion.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have been diagnosed with acute pulmonary embolism on the Aquilion One Genesis scan (Toshiba, Medical System, Tokyo, Japan) at the Brest University Hospital, and who have had a mapping of the iodine derived from the subtraction images.

Exclusion Criteria:

* Tomoscintigraphy not feasible within 24 hours.
* Massive pulmonary embolism or with signs of gravity
* Pregnant or lactating women
* Minor patient
* Protected adults
* Incapacity / refusal to give consent
* Hypersensitivity to pertechnetate (99m Tc)
* Hypersensitivity to human albumin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
The sensitivity of iodine mapping by subtraction technique. | 24 hours
  The sensitivity of iodine mapping by subtraction technique for the detection of perfusion defects in pulmonary embolism is evaluated with using pulmonary perfusion tomoscintigraphy as a reference standard .

SECONDARY OUTCOMES:
The specificity of iodine mapping by subtraction technique | 24 hours
  The specificity of iodine mapping by subtraction technique for the detection of perfusional defects in acute pulmonary embolism is determinated with using pulmonary perfusion tomoscintigraphy as reference standard.
Pulmonary vascular obstruction index | 24 hours
  Thé correlation between the pulmonary vascular obstruction index measured by iodine mapping by subtraction technique and that obtained by perfusion tomoscintigraphy is evaluating
Concordance CTPA - iodine substraction | 24 hours
  The concordance between the morphological abnormalities visualized at the thoracic angioscanner (visualization of an endoluminal defect within the pulmonary arterial network) is evaluated.
Concordance CTPA - SPECT | 24 hours
  The concordance between the morphological abnormalities on CTPA (visualization of an endoluminal defect within the pulmonary arterial network) is evaluated.
Interobserver reproductibility | 24 hours
  The interobserver reproducibility of subtraction technique versus pulmonary tomoscintigraphy in reported as normal or abnormal lung perfusion at a segmental level.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dissaux B, Le Floch PY, Robin P, Bourhis D, Couturaud F, Salaun PY, Nonent M, Le Roux PY. Pulmonary perfusion by iodine subtraction maps CT angiography in acute pulmonary embolism: comparison with pulmonary perfusion SPECT (PASEP trial). Eur Radiol. 2020 Sep;30(9):4857-4864. doi: 10.1007/s00330-020-06836-3. Epub 2020 Apr 11. PMID 32279113